CLINICAL TRIAL: NCT01403311
Title: A Phase 2 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Brief Title: A Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Acronym: ALA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Legacy Health System (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jefferson W Chen, MD, Principal Investigator, Legacy Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5-ALA-01
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Glioma
Keywords: Anaplastic astrocytoma; Astrocytoma; Brain stem glioma; Ependymoma; Glioblastoma; Glioblastoma multiforme; Gliosarcoma; oligodendroglioma; Medulloblastoma; Mixed astrocytoma-ependymoma; ALA
MeSH Terms: conditions — Glioma; Astrocytoma; Ependymoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Medulloblastoma

ARMS (1):
- ALA (Experimental): 5-Aminolevuline Acid (ALA)
  Interventions: Drug: 5-Aminolevuline Acid

INTERVENTIONS:
Drug: 5-Aminolevuline Acid — 5-Aminolevuline Acid (ALA) at 30 mg/kg given orally 4 hours before surgery

SUMMARY:
This study aims to determine the safety and utility of using 5-Aminolevulinic Acid (ALA) in removing malignant brain tumors during surgery.

DETAILED DESCRIPTION:
This study aims to determine the safety and utility of using 5-Aminolevulinic Acid (ALA) in removing brain tumors during surgery. When ALA is provided at an increased concentration, protoporphorin concentration in the malignant cell increases and renders the cell fluorescent under long ultraviolet light. This study looks at using oral ALA to help identify the tumor cells intraoperatively and facilitate complete resection.

Oral ALA will be given prior to image-guided microsurgical resection of the tumor. Following tumor resection under light microscopy, the tumor bed will be illuminated and any residual fluorescent tissue in cavity will be surgically removed leading to a more complete resection of tumor. Pathologic confirmation of tumor type will be made by neuropathology. Photosensitizer concentration in malignant and normal tissue will be estimated by fluorescence microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented primary brain tumor for which resection is clinically indicated. The anticipated histology at resection should include: Anaplastic astrocytoma, Astrocytoma, Brain stem glioma, Ependymoma, Glioblastoma, Glioblastoma multiforme, Gliosarcoma, oligodendroglioma, Medulloblastoma, Mixed astrocytoma-ependymoma
* Patients may have prior therapy
* 18 years of age
* Male or Female
* Life expectancy is not a consideration for protocol entry
* Patients must have normal organ and marrow function as defined below: Leukocytes >3,000/mL, Absolute neutrophil count >1,500/mL, Platelets >100,000/mL, Total bilirubin within normal institutional limits AST (SGOT)/ALT (SGPT)<2.5 X institutional upper limit of normal, Creatinine within normal institutional limits or Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Confirmation of Glial Tumor
* Gross total resection is the aim of surgery
* Ability to understand and the willingness to sign a written informed consent document or have a parent or guardian with the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Non-Glial tumor i.e. tumor abscess, metastasis, lymphoma, vasculitis
* Tumor with perforating vessels
* Tumor involves critical fiber tracks
* Use of the microsurgical tool monopolar loop
* Subject has preexisting severe deficits concerning language or motor function not resolved with steroids
* Performance Status of less than 60
* Prior therapy is not an exclusion criterion
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic acid (ALA)
* Personal or family history of porphorias
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Establish a safe dose to provide optimal discrimination between normal and malignant tissue for oral ALA administration intraoperatively | participants will be followed while in the hospital and for 12 weeks after surgery

SECONDARY OUTCOMES:
Compare time-to-progression and survival to that in comparable cases performed without the aid of ALA | participants will be followed for 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson Chen, MD, PhD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Health System, Portland, Oregon, United States